CLINICAL TRIAL: NCT01964404
Title: Cannabis, Schizophrenia and Reward: Self-Medication and Agonist Treatment?
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Columbia University (Other); Harvard Medical School (HMS and HSDM) (Other); Massachusetts Institute of Technology (Other); Massachusetts General Hospital (Other); Nathan Kline Institute for Psychiatric Research (Other); University of Vermont (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Mary F. Brunette, MD, Principal Investigator, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: D14061; 1R01DA034699-01A1 (NIH)
Record Dates: First submitted 2013-10-15; First posted 2013-10-17 (Estimated); Results first posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-10

CONDITIONS: Schizophrenia; Dual Diagnosis; Psychotic Disorder; Cannabis Use Disorder
Keywords: Dronabinol; Schizophrenia; Dual Diagnosis; Substance Abuse; Cannabis Use Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Substance-Related Disorders | interventions — nabiximols; Dronabinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Marijuana cigarette and placebo capsule (Experimental): 3-5% tetrahydrocannabinol cannabis cigarette smoked immediately prior to the second functional MRI and a placebo capsule (for dronabinol) by mouth taken approximately 2.75 hours prior to the second functional MRI.
  Interventions: Drug: Marijuana
- Dronabinol and placebo cigarette (Experimental): Dronabinol 15mg 3-5% by mouth taken approximately 2.75 hours prior to the second functional MRI and a placebo cigarette (for marijuana) smoked immediately prior to the second functional MRI.
  Interventions: Drug: Dronabinol
- Placebo cigarette and placebo capsule (Placebo Comparator): Placebo cigarette (for marijuana) smoked immediately prior to the second functional MRI and a placebo capsule (for dronabinol) by mouth taken approximately 2.75 hours prior to the second functional MRI.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Marijuana — Smoked plant with THC
  Other Names: Cannabis
  Arms: Marijuana cigarette and placebo capsule
Drug: Dronabinol — Capsule with THC
  Other Names: Marinol
  Arms: Dronabinol and placebo cigarette
Drug: Placebo — Capsule with no active ingredient
  Arms: Placebo cigarette and placebo capsule

SUMMARY:
In this translational research proposal, based on our formulation, we seek to confirm and expand upon data obtained in our pilot study suggesting that cannabis and the cannabinoid agonist dronabinol, given in low dose to patients with schizophrenia and co-occurring cannabis use disorder, will in fact ameliorate the brain reward circuit dysregulation in these patients and, thereby, provide evidence in support of the role of cannabis as a "self-medication" agent for them.

DETAILED DESCRIPTION:
Substance use disorders are strikingly common in patients with schizophrenia and contribute to its morbidity and cost to society. We have proposed a neurobiological formulation suggesting that cannabis and other substance use in these patients may ameliorate a dysfunction in the brain reward circuit(thus serving a "self-medication" function), while also worsening the symptoms and course of schizophrenia.

In this translational research proposal, based on our formulation, we seek to confirm and expand upon data obtained in our pilot study suggesting that cannabis and the cannabinoid agonist dronabinol, given in low dose to patients with schizophrenia and co-occurring cannabis use disorder, will in fact ameliorate the brain reward circuit dysregulation in these patients and, thereby, provide evidence in support of the role of cannabis as a "self-medication" agent for them. Also, by also testing the full range of effects produced by dronabinol (effects on brain reward circuitry assessed with task-based function MRI and resting state connectivity), as well as on reward responsiveness, mood, craving, cognition, psychiatric and extrapyramidal symptoms), we will provide clues as to whether dronabinol should be tried in low doses as an adjunctive agent (with an antipsychotic medication) to limit cannabis use in patients with schizophrenia.

This study will involve 8 groups of 25 participants each. Groups 1-3 will have diagnoses of schizophrenia and cannabis use disorder; Group 4 will have schizophrenia only, Groups 5-7 will have cannabis use disorder only and Group 8 will be healthy control participants. Following screening and baseline neuropsychiatric testing, participants will have two tests days (T1 and T2) that will include task-based functional MRI, including assessment of resting state connectivity, and measuring a number of other parameters including reward responsiveness, mood, craving, symptoms and cognition. The assessments at T1 will be virtually the same for all groups. At T2 Groups 1-3, and Groups 5-7 will be randomly assigned to one of the following conditions prior to the assessments: receiving 15mg of dronabinol and smoking a placebo marijuana cigarette, receiving a placebo pill and smoking a real marijuana cigarette, or receiving a placebo pill and smoking a placebo marijuana cigarette. Group 4 and Group 8 will receive no drug or placebo at T2. Participants receiving drug will have safety assessments before the drug is administered, after the drug is administered but before leaving the research clinic for the day, and again a week later.

ELIGIBILITY:
Inclusion Criteria:

Groups 1-3 Participants with schizophrenia and a cannabis use disorder

1. Ages 18 - 55 years
2. Diagnosis of schizophrenia
3. Diagnosis of cannabis abuse or dependence
4. Use of cannabis within the month prior to screening
5. Willing to remain abstinent for the 14 days before the baseline assessments and throughout the two scans.
6. Psychiatrically stable
7. Treated with a stable dose of an antipsychotic medication (except clozapine) for the past month
8. Not seeking treatment for their cannabis use disorder.

Group 4 - Control participants with schizophrenia

1. Ages 18 - 55 years
2. Diagnosis of schizophrenia
3. Willing to remain abstinent as described above
4. Psychiatrically stable
5. Treated with a stable dose of an antipsychotic medication (except clozapine) for the past month

Groups 5-7 - Control participants with cannabis use disorder

1. Ages 18 - 55 years
2. Diagnosis of cannabis abuse or dependence
3. Use of cannabis within the month prior to screening
4. Willing to remain abstinent as described above
5. Not seeking treatment for their cannabis use disorder.

Group 8 - Healthy control participants

1. Ages 18 - 55 years
2. Willing to remain abstinent as described above

Exclusion criteria:

Groups 1-3 with schizophrenia and a cannabis use disorder

1. Positive symptoms of psychosis (> 4 [moderate]) on any item of the Positive and Negative Syndrome Scale psychosis subscale (once abstinent) except for the hallucination item. We will exclude for a rating > 5 for this item.
2. Cocaine/stimulant use disorder
3. Pharmacological treatment for addiction
4. Mental retardation
5. History of head injury
6. Metal objects within the body that would contraindicate and MRI
7. Pregnancy or currently nursing
8. Uncontrolled medical condition
9. Taking clozapine
10. Any condition that would contraindicate use of cannabis or dronabinol.
11. History of a seizure disorder

Group 4 - Control participants with schizophrenia

1. Positive symptoms of psychosis (> 4 [moderate]) on any item of the Positive and Negative Syndrome Scale psychosis subscale (once abstinent) except for the hallucination item. We will exclude for a rating > 5 for this item.
2. Any history of a substance use disorder other than nicotine
3. Pharmacological treatment for addiction
4. Mental retardation
5. History of head injury
6. Metal objects within the body that would contraindicate and MRI
7. Pregnancy or currently nursing
8. Uncontrolled medical condition
9. Taking clozapine

Groups 5-7 - Control participants with cannabis use disorder

1. Axis I psychiatric diagnosis other than a cannabis use disorder
2. Taking any psychotropic medication
3. Pharmacological treatment for addiction
4. Mental retardation
5. History of head injury
6. Metal objects within the body that would contraindicate and MRI
7. Pregnancy or currently nursing
8. Uncontrolled medical condition
9. History of a seizure disorder

Group 8 - Healthy control participants

1. Any Axis I psychiatric diagnosis
2. Taking any psychotropic medication
3. Pharmacological treatment for addiction
4. Mental retardation
5. History of head injury
6. Metal objects within the body that would contraindicate and MRI
7. Pregnancy or currently nursing
8. Uncontrolled medical condition
9. Current tobacco smokers

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 263 (Actual)
Dates: Start 2014-07; Primary Completion 2021-09-18 (Actual); Study Completion 2021-09-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary F Brunette, MD, Principal Investigator — Dartmouth College
Locations (2):
- United States (2):
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - University of Vermont, Burlington, Vermont

RESULTS

PARTICIPANT FLOW:
Groups:
- Cannabis Use Disorder: Participants met criteria for Cannabis Use Disorder (CUD)
- Dual Diagnosis (Schizophrenia and Cannabis Use Disorder): Participants with a Dual Diagnosis of Schizophrenia and Cannabis Use Disorder
- Schizophrenia: Participants diagnosed with Schizophrenia
- Healthy Controls: Participants with no mental health diagnosis or cannabis use
- Marijuana Cigarette and Placebo Capsule CUD Only: Participants with Cannabis Use Disorder (CUD) and randomized to receive Marijuana Cigarette and Placebo Capsule
- Dronabinol and Placebo Cigarette CUD Only: Participants met criteria for Cannabis Use Disorder (CUD) and were randomized to Dronabinol and Placebo Cigarette
- Placebo Cigarette and Placebo Capsule CUD Only: Participants with a diagnosis of Cannabis Use Disorder (CUD) randomized to Placebo Dronabinol and Placebo Cigarette
- Marijuana Cigarette and Placebo Capsule - SCZ-CUD: Participants with Dual Diagnosis of Schizophrenia and Cannabis Use Disorder (SCZ-CUD) and randomized to Marijuana Cigarette and Placebo Capsule - SCZ-CUD
- Dronabinol and Placebo Cigarette - SCZ-CUD: Participants diagnosed with Diagnosis Schizophrenia and Cannabis Use Disorder and randomized to Dronabinol and Placebo Cigarette
- Placebo Cigarette and Placebo Capsule - SCZ-CUD: Participants diagnosed with Schizophrenia and Cannabis Use Disorder and randomized to placebo Cigarette and Placebo Capsule
Period: Pre-Randomization - Scan 1
Arm/Group | Cannabis Use Disorder | Dual Diagnosis (Schizophrenia and Cannabis Use Disorder) | Schizophrenia | Healthy Controls | Marijuana Cigarette and Placebo Capsule CUD Only | Dronabinol and Placebo Cigarette CUD Only | Placebo Cigarette and Placebo Capsule CUD Only | Marijuana Cigarette and Placebo Capsule - SCZ-CUD | Dronabinol and Placebo Cigarette - SCZ-CUD | Placebo Cigarette and Placebo Capsule - SCZ-CUD
Started (Consented and Screened) | 111 | 79 | 33 | 40 | 0 | 0 | 0 | 0 | 0 | 0
Enrolled and Completed Neuropsych Testing | 62 | 43 | 21 | 31 | 0 | 0 | 0 | 0 | 0 | 0
Completed Scan 1 | 54 | 35 | 18 | 28 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 51 | 34 | 18 | 27 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 60 | 45 | 15 | 13 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Screen Fail | 49 | 36 | 12 | 9 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 8 | 8 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Randomization - Scan 2
Arm/Group | Cannabis Use Disorder | Dual Diagnosis (Schizophrenia and Cannabis Use Disorder) | Schizophrenia | Healthy Controls | Marijuana Cigarette and Placebo Capsule CUD Only | Dronabinol and Placebo Cigarette CUD Only | Placebo Cigarette and Placebo Capsule CUD Only | Marijuana Cigarette and Placebo Capsule - SCZ-CUD | Dronabinol and Placebo Cigarette - SCZ-CUD | Placebo Cigarette and Placebo Capsule - SCZ-CUD
Started (Randomized) | 0 | 0 | 18 | 27 | 17 | 17 | 17 | 11 | 12 | 11
Completed (Completed Scan 2) | 0 | 0 | 18 | 27 | 17 | 17 | 17 | 11 | 12 | 11
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The baseline data includes all participants who were enrolled and completed Neuropsych Testing. Groups have been partitioned to reflect individuals who completed Period 1 (Pre-Randomization -Scan 1) and Period 2 (Randomization- Scan 2)
Groups:
- Marijuana Cigarette and Placebo Capsule SCZ-CUD: 3-5% tetrahydrocannabinol cannabis cigarette smoked immediately prior to the second functional MRI and a placebo capsule (for dronabinol) by mouth taken approximately 2.75 hours prior to the second functional MRI.
  Marijuana: Smoked plant with THC
- Dronabinol and Placebo Cigarette SCZ-CUD: Dronabinol 15mg 3-5% by mouth taken approximately 2.75 hours prior to the second functional MRI and a placebo cigarette (for marijuana) smoked immediately prior to the second functional MRI.
  Dronabinol: Capsule with THC
- Placebo Cigarette and Placebo Capsule. SCZ-CUD: Placebo cigarette (for marijuana) smoked immediately prior to the second functional MRI and a placebo capsule (for dronabinol) by mouth taken approximately 2.75 hours prior to the second functional MRI.
  Placebo: Capsule with no active ingredient
- SCZ-CUD Not Randomized: Dual diagnosis of Schizophrenia and Cannabis Use disorder, - Completed Scan 1 but not Randomized
- Marijuana Cigarette and Placebo Capsule CUD Only: CUD only 3-5% tetrahydrocannabinol cannabis cigarette smoked immediately prior to the second functional MRI and a placebo capsule (for dronabinol) by mouth taken approximately 2.75 hours prior to the second functional MRI.
  Marijuana: Smoked plant
- Dronabinol and Placebo Cigarette CUD Only: CUD only Dronabinol 15mg 3-5% by mouth taken approximately 2.75 hours prior to the second functional MRI and a placebo cigarette (for marijuana) smoked immediately prior to the second functional MRI.
- Placebo Cigarette and Placebo Capsule CUD Only: CUD only Placebo cigarette (for marijuana) smoked immediately prior to the second functional MRI and a placebo capsule (for dronabinol) by mouth taken approximately 2.75 hours prior to the second functional MRI.
- Cannabis Use Disorder - CUD Did Not Randomize: Cannabis Use Disorder (CUD), Completed Scan 1 but not Randomized
- SCZ Only; Healthy Control -: No drug intervention - Completed Scan 1 and 2
- SCZ Only - Did Not Complete Scan 2; Healthy Control - Did Not Complete Scan 2: No drug intervention - Completed Scan 1 but not Scan 2
- Total: Total of all reporting groups
Arm/Group | Marijuana Cigarette and Placebo Capsule SCZ-CUD | Dronabinol and Placebo Cigarette SCZ-CUD | Placebo Cigarette and Placebo Capsule. SCZ-CUD | SCZ-CUD Not Randomized | Marijuana Cigarette and Placebo Capsule CUD Only | Dronabinol and Placebo Cigarette CUD Only | Placebo Cigarette and Placebo Capsule CUD Only | Cannabis Use Disorder - CUD Did Not Randomize | SCZ Only | SCZ Only - Did Not Complete Scan 2 | Healthy Control - | Healthy Control - Did Not Complete Scan 2 | Total
Number analyzed (Participants) | 11 | 12 | 11 | 8 | 17 | 17 | 17 | 10 | 18 | 3 | 27 | 4 | 155
Age, Continuous [Mean (Full Range); unit: Years] | 33.00 [20 to 45] | 28.42 [21 to 46] | 31.55 [21 to 45] | 26.75 [21 to 32] | 43.59 [18 to 54] | 34.29 [20 to 49] | 31.53 [18 to 46] | 34.10 [19 to 48] | 35.55 [19 to 55] | 29.66 [18 to 44] | 33.48 [22 to 53] | 26.5 [18 to 37] | 32.59 [18 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 1 | 3 | 3 | 2 | 2 | 1 | 7 | 1 | 8 | 2 | 35
  Male | 9 | 9 | 10 | 5 | 14 | 15 | 15 | 9 | 11 | 2 | 19 | 2 | 120
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3
  Not Hispanic or Latino | 11 | 11 | 10 | 8 | 17 | 16 | 17 | 10 | 18 | 3 | 27 | 4 | 152
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 3 | 1 | 7
  Black or African American | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 6
  White | 9 | 10 | 9 | 8 | 16 | 15 | 15 | 7 | 17 | 3 | 23 | 3 | 135
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 4
Education, years [Mean (Standard Deviation); unit: Years] | 12.45 (1.695) | 13.92 (1.782) | 13.82 (1.722) | 12.75 (1.165) | 14.12 (1.764) | 14.35 (2.548) | 14.35 (1.967) | 12.8 (1.033) | 13.33 (1.847) | 12 (1) | 17.19 (1.777) | 14.67 (1.155) | 14.28 (2.304)
Schizophrenia, schizoaffective diagnosis [Number; unit: participants]
  Schizophrenia disorder | 3 | 4 | 4 | 6 | 0 | 0 | 0 | 0 | 9 | 1 | 0 | 0 | 27
  Schizoaffective disorder | 8 | 8 | 7 | 2 | 0 | 0 | 0 | 0 | 9 | 2 | 0 | 0 | 36
PANSS [Mean (Standard Deviation); unit: units on a scale] — Positive and Negative Syndrome Scale; Range 7-49, higher score = higher levels of symptoms Population: Measure only collected for subjects with SCZ and SCZ-CUD
  units on a scale
    Positive: number analyzed (Participants) | 11 | 12 | 11 | 8 | 0 | 0 | 0 | 0 | 18 | 3 | 0 | 0 | 63
    Positive | 12.09 (3.91) | 12.83 (3.74) | 12.82 (3.34) | 15.88 (4.88) |  |  |  |  | 13.11 (3.31) | 15.0 (2.65) |  |  | 13.01 (3.73)
    Negative: number analyzed (Participants) | 11 | 12 | 11 | 8 | 0 | 0 | 0 | 0 | 18 | 3 | 0 | 0 | 63
    Negative | 15.82 (8.34) | 12.0 (4.41) | 15.09 (7.91) | 13.63 (3.54) |  |  |  |  | 14.61 (3.96) | 17.66 (6.81) |  |  | 14.19 (5.6)
Days of Cannabis Use in Past 35 [Mean (Standard Deviation); unit: Days] — Days of cannabis use in past 35, range 0-35 days possible
  Days | 10.73 (9.30) | 16.92 (10.10) | 16.64 (10.96) | 18.25 (14.76) | 29.76 (10.14) | 25.18 (12.86) | 24.24 (11.55) | 28.2 (10.35) | 0 (0) | 0 (0) | 0.037 (0.192) | 0.5 (1) | 14.85 (15.54)
Number of Joints Smoked in Past 35 days [Mean (Standard Deviation); unit: Number of Joints] | 18.41 (26.99) | 22.19 (18.82) | 19.70 (16.01) | 44.09 (62.20) | 39.4 (45.3) | 52.2 (78.6) | 52.2 (57.5) | 44.8 (51.2) | 0 (0) | 0 (0) | 0.0357 (0.188) | 0.333 (0.577) | 26.01 (43.45)

OUTCOME MEASURES:

1. Primary Outcome: Brain Reward Circuit Activation on fMRI Scan
Description: Activation of the Brain Reward Circuit (particularly the nucleus accumbens) in anticipation of monetary reward. The 'Measure' is a mean of the Fisher-Z transform of the inter-regional correlation measured for each participant between the nucleus accumbens and anterior cingulate cortex. The Fisher-transformation creates a normally distributed correlation value for statistical analyses assessing between group differences. A Fisher-Z transform of '0' represents a value of '0' for the estimated correlation, which represents no correlation in the activity time series between the regions. The values reflect strengths of functional connectivity between brain regions that can be compared between groups (e.g. Healthy controls and SCZ-CUD groups who received different study drugs). Means and standard deviations similar to healthy controls would be considered a good outcome.
Time Frame: 3 hours
Measure: Mean (Standard Deviation); unit: z-score
Groups:
- Dronabinol and placebo cigarette. SCZ-CUD; Dronabinol and placebo cigarette CUD only: Dronabinol 15mg 3-5% by mouth taken approximately 2.75 hours prior to the second functional MRI and a placebo cigarette (for marijuana) smoked immediately prior to the second functional MRI.
  Dronabinol: Capsule with THC
- Marijuana cigarette and placebo capsule CUD only: 3-5% tetrahydrocannabinol cannabis cigarette smoked immediately prior to the second functional MRI and a placebo capsule (for dronabinol) by mouth taken approximately 2.75 hours prior to the second functional MRI.
  Marijuana: Smoked plant with THC
- Placebo cigarette and placebo capsule. CUD only: Placebo cigarette (for marijuana) smoked immediately prior to the second functional MRI and a placebo capsule (for dronabinol) by mouth taken approximately 2.75 hours prior to the second functional MRI.
  Placebo: Capsule with no active ingredient
- SCZ only: This group of subjects did not have CUD and received no intervention
- Healthy Controls: This group of healthy subjects had no illness and received no intervention
Arm/Group | Marijuana cigarette and placebo capsule SCZ-CUD | Dronabinol and placebo cigarette. SCZ-CUD | Placebo cigarette and placebo capsule. SCZ-CUD | Marijuana cigarette and placebo capsule CUD only | Dronabinol and placebo cigarette CUD only | Placebo cigarette and placebo capsule. CUD only | SCZ only | Healthy Controls
Number analyzed (Participants) | 11 | 12 | 11 | 18 | 17 | 17 | 17 | 27
z-score | 0.05 (0.098) | 0.14 (0.076) | 0.18 (0.127) | 0.12 (0.058) | 0.10 (0.087) | 0.11 (0.081) | 0.17 (0.094) | 0.17 (0.121)
Statistical Analysis 1: Comparison: Marijuana cigarette and placebo capsule SCZ-CUD vs Placebo cigarette and placebo capsule. SCZ-CUD; Test type: Superiority; p = 0.87, t-test, 2 sided — p-FDR; Mean Difference (Final Values) = -0.13

2. Primary Outcome: Resting State Connectivity Within the Brain Reward Circuitry
Description: Resting state connectivity within brain reward circuitry as measured with the Fisher-transformed r value of the connectivity maps between the nucleus accumbans and other brain areas. The Fisher-transformation creates a normally distributed correlation value for statistical analyses assessing between group differences (smoked THC vs placebo; oral dronabinol vs placebo)
Time Frame: 1 hour after smoking study drug, 3 hours after oral dronabinol
Population: Data was collected but cannot be compiled and analysis could not be completed due to death of PI and resulting limited resources for scan data compilation and analyses. There are no immediate resources for analysis in the future.
Arm/Group | Marijuana cigarette and placebo capsule SCZ-CUD | Dronabinol and placebo cigarette. SCZ-CUD | Placebo cigarette and placebo capsule. SCZ-CUD | Marijuana cigarette and placebo capsule CUD only | Dronabinol and placebo cigarette CUD only | Placebo cigarette and placebo capsule. CUD only | SCZ only | Healthy Controls
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: PANSS Positive Symptoms
Description: Positive and Negative Symptom Scale (PANSS) Positive Symptom Mean Subscale Score at 2nd Assessment Day, range 7-49, higher = more symptoms. The outcome measure was recorded at single time of measurement. The time frame includes 3 hours after oral THC/placebo and 1 hour after smoked THC/placebo (the three-hour window is inclusive of the one-hour post smoke). Each individual smoked THC or placebo AND took oral THC or placebo.
Time Frame: 3 hours after oral THC/placebo
Population: Only participants with Schizophrenia were assessed using the Positive and Negative Symptom Scale, as specified in the Study Protocol
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Marijuana cigarette and placebo capsule SCZ-CUD | Dronabinol and placebo cigarette. SCZ-CUD | Placebo cigarette and placebo capsule. SCZ-CUD | SCZ only
Number analyzed (Participants) | 11 | 12 | 11 | 18
score on a scale | 11.0 (0.54) | 9.3 (0.40) | 10.2 (0.56) | 10.6 (0.37)
Statistical Analysis 1: Comparison: Marijuana cigarette and placebo capsule SCZ-CUD vs Placebo cigarette and placebo capsule. SCZ-CUD vs SCZ only; This analysis tested whether the marijuana cigarette group had different PANSS Positive symptom scores compared to the placebo group adjusting for the SCZ only group. (The dronabinol group was tested separately per our analytic plan.); Test type: Superiority; p = 0.31, ANOVA; Mean Difference (Final Values) = 0.82, 95% CI 2-sided [-0.77 to 2.4], Standard Error of Mean 0.81
Statistical Analysis 2: Comparison: Dronabinol and placebo cigarette. SCZ-CUD vs Placebo cigarette and placebo capsule. SCZ-CUD vs SCZ only; This analysis tested whether the dronabinol group had different PANSS Positive symptom scores compared to the placebo group adjusting for the SCZ only group. (The marijuana cigarette group was tested separately per our analytic plan.); Test type: Superiority; p = .62, ANOVA; Mean Difference (Final Values) = -1.2, 95% CI 2-sided [-2.4 to 0.18], Standard Error of Mean .62

4. Secondary Outcome: PANSS Negative Symptoms
Description: Positive and Negative Symptom Scale Negative Symptom Mean Subscale Score at 2nd Assessment Day, range 7-49, higher = more symptoms. The time frame includes 3 hours after oral THC/placebo and 1 hour after smoked THC/placebo (the three-hour window is inclusive of the one-hour post smoke). Each individual smoked THC or placebo AND took oral THC or placebo.
Time Frame: 3 hours after oral THC/placebo
Population: This analysis tested whether the marijuana cigarette group had different PANSS negative symptom scores compared to the placebo group adjusting for the SCZ only group. (The dronabinol group was tested separately per our analytic plan.). Only participants with Schizophrenia were assessed using the Positive and Negative Symptom Scale, as specified in the Study Protocol.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Marijuana cigarette and placebo capsule SCZ-CUD | Dronabinol and placebo cigarette. SCZ-CUD | Placebo cigarette and placebo capsule. SCZ-CUD | SCZ only
Number analyzed (Participants) | 9 | 12 | 11 | 18
score on a scale | 17.1 (0.76) | 16.4 (0.67) | 15.8 (0.81) | 15.2 (0.56)
Statistical Analysis 1: Comparison: Marijuana cigarette and placebo capsule SCZ-CUD vs Placebo cigarette and placebo capsule. SCZ-CUD vs SCZ only; This analysis tested whether the marijuana cigarette group had different PANSS Negative symptom scores compared to the placebo group adjusting for the SCZ only group. (The dronabinol group was tested separately per our analytic plan.); Test type: Superiority; p = 0.28, ANOVA; Mean Difference (Final Values) = 1.2, 95% CI 2-sided [-1 to 3.45]
Statistical Analysis 2: Comparison: Dronabinol and placebo cigarette. SCZ-CUD vs Placebo cigarette and placebo capsule. SCZ-CUD vs SCZ only; This analysis tested whether the dronabinol group had different PANSS Positive negative scores compared to the placebo group adjusting for the SCZ only group. (The dronabinol group was tested separately per our analytic plan.); Test type: Superiority; p = 0.39, ANOVA; Mean Difference (Final Values) = 0.88, 95% CI 2-sided [-1.1 to 2.85], Standard Error of Mean 1.0

5. Secondary Outcome: Cognitive Functioning, Verbal Learning
Description: Cognitive functioning, verbal learning Hopkins Verbal Learning Test (HVLT-R) total raw score. Possible range of scores is 0-35, higher is better functioning. The time frame includes 4 hours after oral THC/placebo and 2 hour after smoked THC/placebo (the three-hour window is inclusive of the one-hour post smoke). Each individual smoked THC or placebo AND took oral THC or placebo.
Time Frame: 4 hours after oral drug
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Marijuana cigarette and placebo capsule SCZ-CUD | Dronabinol and placebo cigarette. SCZ-CUD | Placebo cigarette and placebo capsule. SCZ-CUD | Marijuana cigarette and placebo capsule CUD only | Dronabinol and placebo cigarette CUD only | Placebo cigarette and placebo capsule. CUD only | SCZ only | Healthy Controls
Number analyzed (Participants) | 9 | 12 | 11 | 17 | 16 | 16 | 18 | 27
score on a scale | 23.2 (6.8) | 21.8 (6.7) | 25.0 (5.0) | 25.0 (4.97) | 25.3 (6.1) | 27.9 (4.5) | 25.5 (8.6) | 31.0 (3.3)
Statistical Analysis 1: Comparison: Dronabinol and placebo cigarette. SCZ-CUD vs Placebo cigarette and placebo capsule. SCZ-CUD; This analysis tested whether the dronabinol group had different verbal learning scores compared to the placebo group adjusting for the SCZ only group. (The marijuana cigarette group was tested separately per our analytic plan.); Test type: Superiority; p = 0.004, Regression, Linear — We set threshold of p<.01 for statistical significance due to multiple comparisons; Adjusted for pre-drug exposure cognitive functioning; Mean Difference (Final Values) = -9.98, 95% CI 2-sided [-16.06 to -3.18], Standard Error of Mean 3.424

6. Secondary Outcome: Drug Experience, Anxiety
Description: Drug experience ratings of mood and desirability, anxiety rating on a scale of 0-100, higher means more anxiety.
  The time frame includes 3 hours after oral THC/placebo and 1 hour after smoked THC/placebo (the three-hour window is inclusive of the one-hour post smoke). Each individual smoked THC or placebo AND took oral THC or placebo.
Time Frame: 3 hours after taking oral drug
Population: Only participants with Schizophrenia and CUD who were given study drug were analyzed for drug experiences, as specified in the Study Protocol
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Marijuana cigarette and placebo capsule SCZ-CUD | Dronabinol and placebo cigarette. SCZ-CUD | Placebo cigarette and placebo capsule. SCZ-CUD | SCZ only
Number analyzed (Participants) | 10 | 12 | 11 | 18
units on a scale | 10.03 (4.64) | 3.88 (2.06) | 3.96 (2.30) | 14.31 (4.72)
Statistical Analysis 1: Comparison: Marijuana cigarette and placebo capsule SCZ-CUD vs Placebo cigarette and placebo capsule. SCZ-CUD vs SCZ only; This analysis tested whether the marijuana cigarette group had different anxiety scores compared to the placebo group adjusting for the SCZ only group. (The dronabinol group was tested separately per our analytic plan.); Test type: Superiority; p = .22, Regression, Linear; Mean Difference (Final Values) = 6.07, 95% CI 2-sided [-3.62 to 15.75], Standard Error of Mean 4.94
Statistical Analysis 2: Comparison: Dronabinol and placebo cigarette. SCZ-CUD vs Placebo cigarette and placebo capsule. SCZ-CUD vs SCZ only; This analysis tested whether the dronabinol group had different anxiety scores compared to the placebo group adjusting for the SCZ only group. (The dronabinol group was tested separately per our analytic plan.); Test type: Superiority; p = 0.98, Regression, Linear; Mean Difference (Final Values) = -.88, 95% CI 2-sided [-5.87 to 5.70], Standard Error of Mean 2.95

7. Secondary Outcome: Drug Experience Ratings of Drug Liking
Description: Drug experience ratings of liking rating on a scale of 0-100, higher number = more liking
  The time frame includes 3 hours after oral THC/placebo and 1 hour after smoked THC/placebo (the three-hour window is inclusive of the one-hour post smoke). Each individual smoked THC or placebo AND took oral THC or placebo.
Time Frame: 3 hours after taking oral drug
Population: as for outcome 6
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Marijuana cigarette and placebo capsule SCZ-CUD | Dronabinol and placebo cigarette. SCZ-CUD | Placebo cigarette and placebo capsule. SCZ-CUD
Number analyzed (Participants) | 10 | 12 | 11
units on a scale | 56.5 (21.66) | 56.36 (20.10) | 5.54 (3.49)
Statistical Analysis 1: Comparison: Dronabinol and placebo cigarette. SCZ-CUD vs Placebo cigarette and placebo capsule. SCZ-CUD; This analysis tested whether the dronabinol group had different drug experience ratings of liking scores compared to the placebo group. (The marijuana cigarette group was tested separately per our analytic plan.); Test type: Superiority; p = 0.13, ANOVA; Mean Difference (Final Values) = 50.91, 95% CI 2-sided [10.9 to 90.9], Standard Error of Mean 20.4
Statistical Analysis 2: Comparison: Marijuana cigarette and placebo capsule SCZ-CUD vs Placebo cigarette and placebo capsule. SCZ-CUD; This analysis tested whether the marijuana cigarette group had different drug liking scores compared to the placebo group. (The dronabinol group was tested separately per our analytic plan.); Test type: Superiority; p = .002, Regression, Linear; Mean Difference (Final Values) = 51.1, 95% CI 2-sided [8.01 to 94.07], Standard Error of Mean 21.95

8. Secondary Outcome: Cognitive Function, CPT-IP 2 Digit
Description: Cognitive function, CPT-IP 2 digit measure of Attention. The Continuous Performance Test-Identical Pairs version (CPT-IP)80 assessed attention with range of 1-5, hirer scores indicating better function
  The outcome measure was recorded at single time of measurement. The time frame includes 4 hours after oral THC/placebo and 2 hour after smoked THC/placebo (the three-hour window is inclusive of the one-hour post smoke). Each individual smoked THC or placebo AND took oral THC or placebo.
Time Frame: 4 hours after oral drug
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Marijuana cigarette and placebo capsule SCZ-CUD | Dronabinol and placebo cigarette SCZ-CUD | Placebo cigarette and placebo capsule. SCZ-CUD | Marijuana cigarette and placebo capsule CUD only | Dronabinol and placebo cigarette CUD only | Placebo cigarette and placebo capsule CUD only | SCZ only | Healthy Control -
Number analyzed (Participants) | 11 | 12 | 11 | 17 | 17 | 17 | 18 | 27
score on a scale | 3.5 (0.7) | 3.3 (0.9) | 3.7 (0.7) | 4.1 (0.4) | 3.8 (0.5) | 3.9 (0.4) | 3.2 (1.0) | 4.0 (0.3)
Statistical Analysis 1: Comparison: Dronabinol and placebo cigarette SCZ-CUD vs Placebo cigarette and placebo capsule. SCZ-CUD; Test type: Superiority; p = 0.002, Regression, Linear; Mean Difference (Final Values) = -0.43, 95% CI 2-sided [-1.0 to -0.23], Standard Error of Mean 0.178

ADVERSE EVENTS:
Time Frame: Since past assessment (1-2 weeks)
Arm/Group | Marijuana cigarette and placebo capsule SCZ-CUD | Dronabinol and placebo cigarette SCZ-CUD | Placebo cigarette and placebo capsule. SCZ-CUD | SCZ-CUD not randomized | Marijuana cigarette and placebo capsule CUD only | Dronabinol and placebo cigarette CUD only | Placebo cigarette and placebo capsule CUD only | Cannabis Use Disorder - CUD Did not randomize | SCZ only | SCZ only - Did not complete Scan 2 | Healthy Control - | Healthy Control - Did not complete Scan 2
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/12 | 0/11 | 0/8 | 0/17 | 0/17 | 0/17 | 0/10 | 0/18 | 0/3 | 0/27 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/11 | 0/12 | 1/11 | 1/8 | 0/17 | 0/17 | 0/17 | 1/10 | 2/18 | 0/3 | 0/27 | 0/4
Other Adverse Events (participants affected / at risk) | 9/11 | 9/12 | 8/11 | 2/8 | 14/17 | 10/17 | 14/17 | 5/10 | 13/18 | 3/3 | 14/27 | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Marijuana cigarette and placebo capsule SCZ-CUD (N=11) | Dronabinol and placebo cigarette SCZ-CUD (N=12) | Placebo cigarette and placebo capsule. SCZ-CUD (N=11) | SCZ-CUD not randomized (N=8) | Marijuana cigarette and placebo capsule CUD only (N=17) | Dronabinol and placebo cigarette CUD only (N=17) | Placebo cigarette and placebo capsule CUD only (N=17) | Cannabis Use Disorder - CUD Did not randomize (N=10) | SCZ only (N=18) | SCZ only - Did not complete Scan 2 (N=3) | Healthy Control - (N=27) | Healthy Control - Did not complete Scan 2 (N=4)
Psychosis (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vyvanse Intoxication (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hallucinations (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest Pain (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Marijuana cigarette and placebo capsule SCZ-CUD (N=11) | Dronabinol and placebo cigarette SCZ-CUD (N=12) | Placebo cigarette and placebo capsule. SCZ-CUD (N=11) | SCZ-CUD not randomized (N=8) | Marijuana cigarette and placebo capsule CUD only (N=17) | Dronabinol and placebo cigarette CUD only (N=17) | Placebo cigarette and placebo capsule CUD only (N=17) | Cannabis Use Disorder - CUD Did not randomize (N=10) | SCZ only (N=18) | SCZ only - Did not complete Scan 2 (N=3) | Healthy Control - (N=27) | Healthy Control - Did not complete Scan 2 (N=4)
Anxiety (Psychiatric disorders) | 3 (3) | 2 (2) | 2 (2) | 0 (0) | 4 (4) | 2 (3) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Hallucinations (Psychiatric disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Increased cannabis withdrawal symptoms (Psychiatric disorders) | 3 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psychiatric symptoms (Psychiatric disorders) | 2 (3) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 6 (6) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
hypertension (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dental Issues (Gastrointestinal disorders) | 1 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — This includes dental caries and endodontal abscess
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety in MRI (Psychiatric disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 2 (2) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back, shoulder or neck pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 4 (8) | 0 (0)
MRI Finding - Nervous System (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 0 (0) | 2 (2) | 0 (0) — Arachnoid cyst, Berry Aneurysm, Leukoencephalopathy, herniation of sella, 1.3 cm cyst, elevated signal hemibrain + pons, benign mass, cystic lesion, lesion, enlargement of pituitary gland, white matter signal abnormality
Chest Pain (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea or vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 1 (3) | 0 (0) — Fall, sprained knee, heel abrasion, bruising at IV insertion site
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 2 (4) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 4 (4) | 0 (0)
Hemorrhoids (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Hemorrhoidectomy
Chalazia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abnormal EKG (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lightheaded/Dizzy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Dysesthesia/Parasthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Foot fungus
Muscle aches (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MRI Findings - Vascular (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MRI Findings - Respiratory (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Swelling of vein (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Other (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Syncope, Tremor, Migraine

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-27): https://cdn.clinicaltrials.gov/large-docs/04/NCT01964404/Prot_SAP_000.pdf